CLINICAL TRIAL: NCT02903706
Title: Prevalence of Malaria Parasites in People Working in Illegal Gold Mining in French Guiana
Acronym: ORPAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: ORPAL
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Malaria; Epidemiology
Keywords: gold miners; plasmodium carriers; artemisinine resistance
MeSH Terms: conditions — Malaria | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample (5 ml) for Plasmodium PCR
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measure of Plasmodium prevalence (PCR)

SUMMARY:
Malaria is the most widespread parasitic illness in the world, and it is endemic to Guiana. Although the number of cases has decreased since 2005, sources of infection still remain, particularly within illegal gold mines. These malaria carriers/sufferers often use self-medication to deal with malaria symptoms, resulting in a risk of resistance to anti-malarial treatments, and particularly to artemisinine. The mobility of this population across the Guiana Shield increases both the risk of malaria spreading and the resistance of this illness to treatment in the region, and puts the population at risk of new outbreaks of this disease despite the great efforts put into anti-malarial policy in this region.

Fighting malaria within this population is therefore a dual public health challenge: on the one hand, make it possible for the WHO to eliminate malaria from the Guiana Shield by 2017, on the other to limit resistance to artemisinine in this region. However, Guiana's particular context - namely the illegal status of gold mines and the difficult geographical access, the Harpie military operations, the illegality of carrying out malarial diagnosis tests and treating cases without the presence of a health professional - prevents us from achieving this goal using the same tools as our neighbours in Suriname, whose " Looking for Gold, Finding Malaria " programme was a success.

A better understanding of the malarial epidemiology in this population will enable us to propose innovative, more adapted measures to combat malaria within these guyanese populations. This is an transversal, multicentric observational study.

DETAILED DESCRIPTION:
Main Aim:

To estimate the prevalence of Plasmodium carriers in the population of illegal gold mine workers in French Guiana.

Secondary aims:

Evaluate the proportion of different Plasmodium species affecting this population and

* Determine parasitaemia levels;
* Evaluate the gametocyte index;
* Map the number and proportion of P. falciparum cases for the different river sites where gold mining is carried out;
* Determine the lifestyle, knowledge, attitude and behaviour of these populations concerning malaria;
* Estimate the prevalence of mutations linked to the resistance of parasites to artemisinine derivatives;
* Analyse the global genetic diversity of these parasites.
* Evaluate the global health of gold miners

The results of this study will make it possible to characterise the malaria epidemic in illegal gold-mining sites across French Guiana, evaluate the size of the human reservoir and the prevalence of ACT-tolerant parasites, identify the most urgent areas to be dealt with, suggest appropriate plans of action for this, and adopt more efficient public information campaigns.

Target Population: People working on illegal gold mining sites in French Guiana.

Inclusion Criteria:

* works on a gold mining site in French Guiana
* has been at the resting site for less than seven days
* is over the age of 18
* accepts to take part in this study

Exclusion Criteria:

* refuses to take part in the study
* is under the age of 18

The sampling of the 240 people needed for this study will be achieved through chance meetings and the resulting snowball effect at gold mining resting sites on the Surinamese banks of the Maroni river.

Study Protocol:

* Acquisition of authorisations from the competent French authorities
* Authorisation from the competent Surinamese authorities
* Recruitment of one mediator/translator, one state registered nurse and one doctor
* Collaboration with Dr Cairo (program "looking for gold, finding malaria) in Suriname to plan the field missions
* Teams from Suriname and French Guiana will work joinly in the field: eligible persons will be enrolled in the study, the others can be tested by the Surinamese team.
* Inclusion of subjects through chance meetings and the snowball effect at resting sites
* Consent of patients and checking of inclusion criteria
* Performance of three diagnostic tests for each person, including

  * an RDT on site
  * If the RDT is positive: complete treatment given to patient following national guidelines;
  * If necessary, provision of a results sheet describing the necessary doses for treatment;

    * Performance of thick and thin blood smears for transport to the CHAR parasitology laboratory for analysis;
    * Collection of a 5ml (EDTA) tube of blood d'un tube de sang de 5ml reserved in an icebox between 4°C et 10°C for the CNR malarial parasitology lab at the Institut Pasteur de la Guyane;
* Completion of the questionnaire;
* Temperature is taken;
* Patient is provided with a brochure about malaria in Portugese and/or Sranantango;
* Provision of an insecticide-treated net.

ELIGIBILITY:
Inclusion Criteria:

* works on a gold mining site in French Guiana
* has been at the resting site for less than seven days
* is over the age of 18
* accepts to take part in this study

Exclusion Criteria:

* refuses to take part in the study
* is under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People working on illegal gold mining sites in French Guiana.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
prevalence of malaria positive individuals (symptomatic or not symptomatic) | 1 month
  every participant gives a capillary blood specimen which is then screened for malaria using PCR in order to obtain a prevalence of malaria positive individuals (symptomatic or not symptomatic)

SECONDARY OUTCOMES:
Microscopy: thick and thin smear | 1 month
  Each participant is screen for malaria using classic microscopy on thin and thick smears in order to obtain a prevalence of malaria positive individuals and to evaluate parasite quantities, and gametocyte carriage (transmission potential). If either thin or thick smears are positive then the patient is estimated to have smear positive malaria.

REFERENCES:
- [Derived] Douine M, Mosnier E, Le Hingrat Q, Charpentier C, Corlin F, Hureau L, Adenis A, Lazrek Y, Niemetsky F, Aucouturier AL, Demar M, Musset L, Nacher M. Illegal gold miners in French Guiana: a neglected population with poor health. BMC Public Health. 2017 Jul 17;18(1):23. doi: 10.1186/s12889-017-4557-4. PMID 28716015